CLINICAL TRIAL: NCT07000253
Title: Timing of Minimally Invasive Local Treatment After First-Line Systemic Therapy in Oligometastatic Esophageal or Gastric Adenocarcinoma: A Randomized Prospective Clinical Study (OMEC-5)
Brief Title: Timing of Minimally Invasive Local Treatment After First-Line Systemic Therapy in Oligometastatic Esophageal or Gastric Adenocarcinoma
Acronym: OMEC-5
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Hanneke W. M. van Laarhoven, prof . dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMEC-5
Record Dates: First submitted 2025-05-08; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer; Gastric (Stomach) Cancer; Gastric Adenocarcinoma; Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma or Esophageal Carcinoma; Esophageal Carcinoma; Gastric (Cardia, Body) Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasms | interventions — Drug Therapy; Immunotherapy; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- long duration of systemic therapy (Experimental): Patients with no disease progression at 4 months (18 weeks) after systemic therapy with oxaliplatin, fluorpyrimidine, checkpoint inhibitor and/or taregted therapy and fit for local treatment will receive 4 additional months of systemic therapy and subsequent evaluation for local treatment to all disease sites.
  Interventions: Drug: Chemotherapy; Drug: Targeted Systemic Therapy; Drug: Immunotherapy; Procedure: Surgery; Radiation: Radiotherapy
- Short duration of systemic therapy (Active Comparator): Patients with no disease progression at 4 months (18 weeks) after systemic therapy oxaliplatin, fluorpyrimidine, checkpoint inhibitor and/or targeted therapy and fit for local treatment will recieve direct local treatment to all disease sites.
  Interventions: Drug: Chemotherapy; Drug: Targeted Systemic Therapy; Drug: Immunotherapy; Procedure: Surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy preferably CapOx (capecitabine + oxaliplatin) or FOLFOX (5-fluoruracil, leucovorin and oxaliplatin) will be combined with immunotherapy (preferably nivolumab or pembrolizumab) and/or targeted therapy (for example trastuzumab in the case of HER2 overexpression or zolbetuximab in the case of Claudin 18.2 overexpression). These regiments are the standard-of-care (SOC) combination therapies used in this study. Acceptable chemotherapy regimens predominantly for Asian centers include SOX (S-1 and Oxaliplatin).
Drug: Targeted Systemic Therapy — Biomarker selected patients will receive trastuzumab, zolbetuximab or any other targeted agent according to standard of care.
Drug: Immunotherapy — Biomarker selected patients will recieve checkpoint inhibitors according to standard care
Procedure: Surgery — If the primary tumor is present, this tumor will be surgically removed. Metastases may also be removed by surgery.
Radiation: Radiotherapy — Metastases may be irradiated

SUMMARY:
Purpose of the Study:

This clinical study investigates whether a shorter or longer duration of systemic therapy before local treatment (surgery or radiation) results in better disease control in patients with esophageal or gastric cancer with a limited number of metastases, also known as oligometastases.

Background:

In about 25% of patients with advanced esophageal or gastric cancer, the disease spreads to only a few sites (oligometastatic disease). Prior studies suggest that local treatment after systemic therapy may extend survival in this subgroup. However, it is unclear how long systemic therapy should last before initiating local treatment. The OMEC-5 study aims to clarify this and identify potential biomarkers for treatment response.

Study Design:

Initiated by Amsterdam UMC and UMCU and conducted in multiple hospitals across Europe.

Total of 414 patients to be enrolled.

Duration: ~53 months (35 months enrollment + 18 months follow-up).

Approved by the medical ethics committee at Amsterdam UMC.

Procedure:

Eligibility screening: Includes physical exam, blood tests (incl. circulating tumor cells), medical history review, and confirmation of oligometastases by an expert panel.

Initial treatment: All participants receive 4 months of standard systemic therapy (chemotherapy + immunotherapy and/or targeted therapy depending on tumor markers like HER2 or Claudin 18.2).

Response assessment (Review 1): Imaging and/or laparoscopic examination.

If oligometastases persist and tumors have not progressed, participants are randomized into two groups:

Group A (longer systemic therapy): 4 more months of systemic therapy, then local treatment if disease is stable, followed by 4 months of immunotherapy ± targeted therapy.

Group B (shorter systemic therapy): Immediate local treatment followed by 4 months of systemic therapy, then reassessment and potentially 4 months of immunotherapy ± targeted therapy.

Follow-up: Regular scans and quality-of-life questionnaires (5 times), and periodic blood sampling (4 times).

Treatments Involved:

Chemotherapy: CapOx or FOLFOX

Immunotherapy: nivolumab or pembrolizumab

Targeted therapy: trastuzumab (HER2-positive) or zolbetuximab (Claudin 18.2-positive)

Potential Benefits and Risks:

Patients may benefit from better disease control and a personalized treatment strategy.

Known side effects relate to the standard treatments used (chemo, immuno, targeted therapies), and no extra medical risk is expected beyond routine care.

Possible inconveniences include blood draws, scans, minor surgery (laparoscopy), and time investment.

Data and Sample Handling:

Personal data and tumor/blood samples are coded and securely stored.

Data may be used for future cancer research if the patient consents.

Participants can withdraw at any time.

Confidentiality and Privacy:

Patient data are kept confidential, and participants have rights to access or delete their data. Privacy measures comply with GDPR and Dutch law.

Compensation and Insurance:

Participation is voluntary, with no financial compensation. Standard treatment costs are covered by healthcare insurance. No extra insurance is required, as the treatment aligns with standard care practices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability to provide written informed consent
* Histologically confirmed esophageal, gastric or gastroesophageal junction tumor with oligometastatic (M1) disease defined according to the OMEC consensus statement:

  * One organ with ≤3 metastases or 1 involved extra-regional lymph node station (based on the TNM 8 classification)
  * ≤3 unilobar liver metastases or ≤2 bilobar liver metastases
  * ≤ 3 unilateral lung metastases
  * Unilateral adrenal gland involvement
  * Metastasis confined to 1 bone structure or 1 soft tissue compartment
* Synchronous oligometastatic disease with a resectable primary tumor or metachronous oligometastatic disease (in the event of a locoregional recurrence this should be resectable)
* Metastases should be deemed amenable by the international multidisciplinary expert team for radical local treatment
* WHO performance status 0-2
* Indication for checkpoint inhibition and/or targeted therapy

  * PD-L1 with a CPS of 1 or higher as per local clinical practice for immunotherapy use
  * HER2 overexpression as per local clinical practice for trastuzumab use
  * Claudin 18.2 overexpression as per local clinical practice for zolbetuximab use.
  * Any other biomarker that allows targeted therapy in first line approved by EMA
* No prior systemic therapy for metastatic disease
* CT-scan ≤8 weeks prior to inclusion
* Ability to undergo local treatment and start systemic treatment beyond 18 weeks of total systemic treatment.

Exclusion Criteria:

* Squamous cell carcinoma
* Brain metastases
* Peritoneal or pleural carcinomatosis
* Patients with MSI dMMR
* Uncontrolled immunodeficiency (e.g. AIDS)
* Peripheral neuropathy >CTCAE grade 1, precluding start of full dose oxaliplatin treatment
* Both organ metastasis and extra-regional lymph node metastasis
* Conditions precluding local treatment or systemic therapy for oligometastatic disease:

  * Serious medical comorbidities precluding local treatment (e.g., interstitial lung disease in patients with pulmonary metastasis)
  * Clinical or radiological evidence of spinal cord compression or epidural tumor within 2 mm of the spinal cord
  * Simultaneous other malignancy or previous other malignancy with a disease-free period of <5 years, except adequately treated non-melanoma skin cancer or in-situ cancers
  * Uncontrolled (bacterial) infections
  * Significant concomitant diseases preventing the safe administration of study drugs or likely to interfere with study assessments
  * Uncontrolled angina pectoris, cardiac failure or clinically significant arrhythmias
  * Continuous use of immunosuppressive agents equivalent to >10 mg daily prednisone
  * Concurrent use of the antiviral agent sorivudine or chemically related analogues, such as brivudine
  * Pregnancy or breast feeding
  * Patients (M/F) with reproductive potential not implementing adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-06 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | the time interval from the date of randomization to the date of first occurrence of the following events (or last follow-up) up to 53 months after study initiation: Disease progression, death
  the time interval from the date of randomization to the date of first occurrence of the following events (or last follow-up) up to 53 months after study initiation:
  * Disease progression (consisting of either progression in the number of metastases, recurrence at surgically treated metastasis, progression of ablated or irradiated metastasis, or recurrence of the primary tumor or regional lymph node metastasis)
  * Death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Interval between randomization and death or last follow-up up to 53 months after study initiation
2. Quality of Life (QoL) | At 12 months after randomization.
  Measured by the Summary Score of the EORTC QLQ-C30

OTHER OUTCOMES:
Levels of ctDNA circulating in plasma | before start of systemic treatment (t=0), at restaging (t=4 months) and during follow-up (at t= 8 months and t = 12 months)
Potential new (blood or tissue based) biomarkers that predict clinical outcome and response to treatment | before start of systemic treatment (t=0), at restaging (t=4 months) and during follow-up (at t= 8 months and t = 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Peter van Rossum, MD, PhD, Principal Investigator — Amsterdam UMC; Richard van Hillgersberg, MD, PhD, Principal Investigator — UMC Utrecht; Hanneke van Laarhoven, MD, PhD, PhD, Principal Investigator — Amsterdam UMC; Tiuri Kroese, MD, PhD, Study Director — University of Zurich
Locations (2):
- Netherlands (2):
  - Amsterdam Univeristy Medical Center, Amsterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Description of the complete OMEC protocol — https://omecprojects.com/